CLINICAL TRIAL: NCT03636399
Title: Group Based Treatment for Persons With Social Communication Difficulties: A Randomized Controlled Trial
Brief Title: Group Based Treatment for Persons With Social Communication Difficulties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Silje Merethe Hansen, Co-Principal Investigator, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1360
Record Dates: First submitted 2018-08-12; First posted 2018-08-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Brain Injuries
Keywords: adults; rehabilitation; social communication disorder; cognitive communication disorder; groups; evidence-based
MeSH Terms: conditions — Brain Injuries; Social Communication Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard GIST (Experimental): Standard Group Interactive Structured Treatment.
  Interventions: Behavioral: Standard GIST
- Waitlist control/Intensive GIST (Other): After a wait list control period of nine months the participants receive Intensive Group Interactive Structured Treatment.
  Interventions: Behavioral: Intensive GIST

INTERVENTIONS:
Behavioral: Standard GIST — 13 group modules will be administered to outpatients in 12 x 2,5-3 hours sessions. Manualized intervention; In every group session a new topic is presented, discussed and practiced in group exercises. Homework assignments between sessions.
  Other Names: GIST
  Arms: Standard GIST
Behavioral: Intensive GIST — 13 group modules will be administered to inpatients during 4 weeks in hospital. Participants is admitted to a hospital unit for cognitive rehabilitation treating patients in acute and/or cronic phase. The participants are given extended leave every weekend to work on homework Assignments between each treatment week.
  Other Names: GIST
  Arms: Waitlist control/Intensive GIST

SUMMARY:
A large proportion of patients with ABI have cognitive deficits that affect the way they communicate. Cognitive difficulties with attention, memory, executive functions and so on affect social communication. Without successful social skills, a person may engage in conflicts, become isolated and be denied access to social and vocational opportunities. Internationally, several group interventions have been developed for treating social communication difficulties during the last years.

Group Interactive Structured Treatment (GIST) is a validated holistic multidisciplinary group treatment targeting social communication skills after traumatic brain injury. The main aim of the present study is to examine the efficacy of GIST for improving social communication in persons with acquired brain injury, including TBI, stroke, tumor ect. Secondary the study aims to compare the standard GIST protocol to an newly developed intensive GIST protocol. Efficacy will be assessed immediately after intervention, but also three and six months after the intervention. The project is in line with international research efforts aimed to establish more knowledge about group treatment for persons with social communication disorders after ABI.

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury (TBI), cerebrovascular accidents (stroke; CVA) patients with no concomitant diseases minimum 6 months post-injury
* The patient are experiencing social communication disorders
* The family member is experiencing the patients social communication disorders
* The patient is motivated and expresses a desire to change communication behavior
* One close family member is able to participate in the intervention process
* Adequate Norwegian language proficiency to participate in the group
* The patient experiences moderate to severe difficulties with minimum 3 aspects of communication assessed with La Trobe Questionnaire
* The patient have insight into their communication difficulties (minimum intellectual insight) assessed with Awareness Questionnaire

Exclusion Criteria:

* Age <18 years
* Aphasia. Based on previous records.
* Major psychiatric disorder or reported ongoing alcohol or substance abuse
* Premorbid neurological disease or insult and/or comorbid neurological disease
* Impaired basic linguistic, mnemonic, motor, or perceptual function that can interfere with the ability to engage with the training or intelligence quotient (IQ) < 85

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
La Trobe Questionnaire. | Change from baseline up to 6 months
  The LaTrobe Communication Questionnaire (LCQ) is a 30-item questionnaire that measures communication ability, a subjective outcome measure. Various communication behaviours are rated on a 4-point scale: 1¼never or rarely, 2¼sometimes, 3¼often and 4¼usually or always, but six items require a reverse in the scoring. Higher scores reflect reduced communications skills. The tool was developed to obtain information from various sources (e.g. self -rating by individual with TBI, rating by support person).

SECONDARY OUTCOMES:
Profile of Pragmatic Impairment in Communication (PPIC) | Change from baseline up to 6 months
  PPIC is an objective measure of social communication skills designed specifically for use with people with TBI. It includes 10 feature summary scales that assess communication skills on a 6-point scale from normative (0) to very severely impaired (5), with lower scores indicating better performance. These summary scales-logical content; general participation; quantity; quality; internal relation; external relation; clarity of expression; social style; subject matter; and aesthetics.
Mind in the eyes test | Change from baseline up to 6 months
  This test consists of 36 black- and-white pictures of the eye region. The images are presented one by one, along with four adjectives (one target word and three foil words).
Goal Attainment Scaling (GAS) | Change from baseline up to 6 months
  Goal Attainment Scaling (GAS) is a flexible system of measuring outcome goals, based on a 5-point scale.
  Levels of goal attainment are expressed objectively in terms of concrete behaviors that can be observed and recorded.
Behavior Rating Inventory for Executive Functions (BRIEF) | Change from baseline up to 6 months
  BRIEF is a 75-item self and other questionnaire that measures executive functions (inhibition, shift, emotional control, self-monitoring, initiative, working memory, planning/organizing, task monitoring, organizing of materials)communication ability. Various executive behaviours are rated on a 3-point scale.
Social competence checklist | Change from baseline up to 6 months
  Is an interview where the participant and close family member answer 6 yes or no answers regarding the participants social communication skills. The interview is found in the GIST protocol developed by Hawley and Newman 2002.
CIQ (Community Integration Questionnaire) | Change from baseline up to 6 months
  The Community Integration Questionnaire (CIQ) is a community integration outcome measure developed for TBI subjects; its social integration and productivity subscales were used for this study. Frequency of such activities as shopping, leisure pursuits, visiting friends or relatives, travel, and one's work, school, or volunteer situation, are scored on a 15-item scale; a higher score indicates greater integration.
Norwegian Version of the General Perceived Self-Efficacy Scale | Change from baseline up to 6 months
  is a 20-item questionnaire that measures self-efficacy rated by a 4-point scale.
Norwegian Quality of Life Scale (PQoL), | Change from baseline up to 6 months
  is a 20-item questionnaire that measures quality of life, a subjective outcome measure. The quality of life is rated in a 0-10 point scale. Higher scores reflect high quality of life.
Symptom Checklist (SCL-10) | Change from baseline up to 6 months
  To document self-reported psychological problems and symptoms of psychopathology, the Symptom Checklist 90-R was used.
Social Communication Questionnaire with additional questions (SCQ-A) | Change from baseline up to 6 months
  SCQ-A is a 37-item questionnaire that measures communication ability, a subjective outcome measure. Various communication behaviours are rated on a 5-point scale. Higher scores reflect reduced communications

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Kirmess, PHD, Principal Investigator — Sunnaas Sykehus
Locations (1):
- Sunnaas rehabilitation hospital, Nesoddtangen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen SM, Stubberud J, Hjertstedt M, Kirmess M. Intensive and standard group-based treatment for persons with social communication difficulties after an acquired brain injury: study protocol for a randomised controlled trial. BMJ Open. 2019 Sep 8;9(9):e029392. doi: 10.1136/bmjopen-2019-029392. PMID 31501112
- [Derived] Ingebretsen SMH, Kirmess M, Smastuen MC, Hawley L, Newman J, Stubberud J. Rehabilitation of Social Communication Skills in Patients With Acquired Brain Injury With Intensive and Standard Group Interactive Structured Treatment: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 Jul;104(7):1016-1025. doi: 10.1016/j.apmr.2023.02.023. Epub 2023 Mar 24. PMID 36966953